CLINICAL TRIAL: NCT00756652
Title: MemoryGel Silicone Gel-Filled Breast Implant Post-Approval Study
Brief Title: Mentor MemoryGel Post-Approval Study
Acronym: MGPAS
Status: Completed | Type: Observational
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P030053; NCT00495534 (obsolete NCT alias)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Breast Reconstruction; Breast Augmentation; Breast Revision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MemoryGel Breast Implant Participants: MemoryGel Breast Implant Participants received Mentor Silicone Gel-Filled Breast Implants (MemoryGel) during their Breast Augmentation, Breast Reconstruction, or Revision surgery
  Interventions: Device: Mentor Silicone Gel-Filled Breast Implants
- Saline Breast Implant Control Participants: Saline Breast Implant Control Participants received Saline Filled Breast Implants during their Breast Augmentation, Breast Reconstruction, or Revision surgery
  Interventions: Device: Saline Breast Implants

INTERVENTIONS:
Device: Mentor Silicone Gel-Filled Breast Implants
  Other Names: MemoryGel Breast Implants
  Groups: MemoryGel Breast Implant Participants
Device: Saline Breast Implants
  Groups: Saline Breast Implant Control Participants

SUMMARY:
In November 2006, U.S. Food and Drug Administration (FDA) approved Mentor's MemoryGel silicone gel-filled breast implants for use in women who are undergoing primary or revisional breast augmentation and primary or revisional breast reconstruction surgery. This postapproval study is intended to satisfy one element of FDA's postapproval monitoring requirements. In January 2015, the FDA approved a protocol amendment that limits the scope of data collection for the study to the collection of only secondary procedure/reoperation data for MemoryGel participants.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 18 years or older (22 or older for breast augmentation patients)
2. U.S. resident

Exclusion Criteria:

1. If a saline participant, current or past, unilateral or bilateral, silicone breast implants
2. Active infection anywhere in her body
3. Existing breast cancer or pre-cancer of the breast without adequate treatment for those conditions
4. Currently pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MemoryGel™ PAS uses a current cohort design of 41,900 gel participants and 1,000 saline participants.
Sampling Method: Non-Probability Sample
Enrollment: 42491 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Canady, M.D., Study Director — Mentor Worldwide, LLC

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In January 2015, the FDA approved a protocol amendment that limited the scope of the study to the collection of only secondary procedure and reoperation data for the MemoryGel arm participants. No data collection is required for the Saline Breast Implant Control group participants and no outcome measures are reported for this study arm.
Groups:
- MemoryGel Breast Implant Participants: Subjects who received Mentor Silicone Gel-Filled Breast Implants (MemoryGel) during their Breast Augmentation, Breast Reconstruction, or Revision surgery
- Saline Breast Implant Control Participants: Subjects who received Saline Filled Breast Implants during their Breast Augmentation, Breast Reconstruction, or Revision surgery
Period: Original Phase
Arm/Group | MemoryGel Breast Implant Participants | Saline Breast Implant Control Participants
Started | 41452 | 1039
Completed | 6063 (At Year 7) | 118
Not Completed | 35389 | 921
Not completed — Withdrawal by Subject | 864 | 23
Not completed — Lost to Follow-up | 601 | 0
Not completed — Other Discontinuation | 797 | 5
Not completed — Participant Noncompliance | 18622 | 424
Not completed — Unknown Discontinuation Reason | 2 | 0
Not completed — Participants without data | 3259 | 466
Not completed — Death | 168 | 1
Not completed — Not due for F/U at Phase One closure | 11076 | 2
Period: Re-Op Phase
Arm/Group | MemoryGel Breast Implant Participants | Saline Breast Implant Control Participants
Started | 11101 | 0 (NA - The Re-Op Phase was limited in scope to data collection for only MemoryGel participants.)
Completed | 8225 | 0
Not Completed | 2876 | 0
Not completed — Withdrawal by Subject | 62 | 0
Not completed — Death | 6 | 0
Not completed — Lost to Follow-up | 340 | 0
Not completed — Site Closed | 2454 | 0
Not completed — Withdrawn after explant | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Original Phase - MemoryGel Participants: Subjects implanted with MemoryGel breast implants
- Original Phase - Saline Breast Implant Control Participants: Subjects implanted with saline filled breast implants
- Total: Total of all reporting groups
Arm/Group | Original Phase - MemoryGel Participants | Original Phase - Saline Breast Implant Control Participants | Total
Number analyzed (Participants) | 41452 | 1039 | 42491
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.3 (11.4) | 32.1 (9.9) | 40.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41452 | 1039 | 42491
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White, not of Hispanic origin | 32216 | 575 | 32791
  White, of Hispanic origin | 4123 | 262 | 4385
  Black, not of Hispanic origin | 891 | 28 | 919
  Black, of Hispanic origin | 146 | 11 | 157
  Asian, Asian American, Pacific Islander | 1873 | 74 | 1947
  Native American or Alaskan Native | 306 | 8 | 314
  Other | 1025 | 44 | 1069
  Missing | 872 | 37 | 909
Surgery Indication [Number; unit: Participants]
  Primary Augmentation | 26173 | 937 | 27110
  Revision Augmentation | 8382 | 75 | 8457
  Primary Reconstruction | 5023 | 15 | 5038
  Revision Reconstruction | 1761 | 9 | 1770
  Unknown Indication | 113 | 3 | 116

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimated Cumulative Incidence of Reported Complications
Description: The KM estimated cumulative incidence of reoperation and explantation has been estimated on a patient-level basis. The data for the KM analysis used the follow-up and reoperation/explantation reports from the entire data set of the 41,452 participants in the Original study, with follow-up and additional reoperartions/explantations reported on the 11,101 participants in the ReOperation phase. Participants with no post-op follow-up are excluded from the KM analysis.
Time Frame: 10 years
Population: Per the FDA-approved protocol amendment, no data collection is required for the Saline Breast Implant Control group participants and no outcome measures are reported for this study arm.
  The number of participants each year is based on participants with post-op follow-up in that year
Measure: Number (95% Confidence Interval); unit: Cumulative Reoperation Events
Groups:
- MemoryGel Participants: Subjects who received MemoryGel breast implants
Arm/Group | MemoryGel Participants
Number analyzed (Participants) | 41452
Cumulative Reoperation Events
  0 Years: number analyzed (Participants) | 11158
  0 Years | 0.0 [0 to 0]
  1 Year: number analyzed (Participants) | 8779
  1 Year | 6.7 [6.2 to 7.2]
  2 Years: number analyzed (Participants) | 4792
  2 Years | 10.8 [10.1 to 11.4]
  3 Years: number analyzed (Participants) | 4613
  3 Years | 11.2 [10.5 to 11.8]
  4 Years: number analyzed (Participants) | 4525
  4 Years | 11.7 [11.0 to 12.4]
  5 Years: number analyzed (Participants) | 4336
  5 Years | 12.5 [11.8 to 13.2]
  6 Years: number analyzed (Participants) | 4228
  6 Years | 13.0 [12.3 to 13.8]
  7 Years: number analyzed (Participants) | 4159
  7 Years | 13.2 [12.5 to 14.0]
  8 Years: number analyzed (Participants) | 4047
  8 Years | 13.3 [12.6 to 14.1]
  9 Years: number analyzed (Participants) | 3910
  9 Years | 13.6 [12.8 to 14.4]
  10 Years: number analyzed (Participants) | 3493
  10 Years | 13.7 [12.9 to 14.5]

2. Primary Outcome: Kaplan Meier Estimated Cumulative Incidence of Explantation
Description: as for outcome 1
Time Frame: 10 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative Explantation Events
Arm/Group | MemoryGel Participants
Number analyzed (Participants) | 41452
Cumulative Explantation Events
  0 Years: number analyzed (Participants) | 11158
  0 Years | 0 [0 to 0]
  1 Year: number analyzed (Participants) | 9037
  1 Year | 3.0 [2.7 to 3.4]
  2 Years: number analyzed (Participants) | 5003
  2 Years | 5.0 [4.6 to 5.5]
  3 Years: number analyzed (Participants) | 4831
  3 Years | 5.2 [4.7 to 5.7]
  4 Years: number analyzed (Participants) | 4752
  4 Years | 5.5 [5.0 to 6.1]
  5 Years: number analyzed (Participants) | 4561
  5 Years | 6.0 [5.4 to 6.5]
  6 Years: number analyzed (Participants) | 4454
  6 Years | 6.4 [5.8 to 6.9]
  7 Years: number analyzed (Participants) | 4386
  7 Years | 6.5 [6.0 to 7.1]
  8 Years: number analyzed (Participants) | 4273
  8 Years | 6.6 [6.1 to 7.2]
  9 Years: number analyzed (Participants) | 4133
  9 Years | 6.8 [6.2 to 7.4]
  10 Years: number analyzed (Participants) | 3698
  10 Years | 6.9 [6.3 to 7.6]

3. Secondary Outcome: Reasons for Reoperations
Description: Frequencies of the reason for reoperation will be computed for women with MemoryGel breast implants through 10 years
Time Frame: 10 Years
Population: In January 2015, the FDA approved a protocol amendment that limited the scope of the study to the collection of only secondary procedure and reoperation data for the MemoryGel arm participants. No data collection is required for the Saline Breast Implant Control group participants and no outcome measures are reported for this study arm.
Measure: Number; unit: Reoperation events
Arm/Group | MemoryGel Participants
Number analyzed (Participants) | 1141
Reoperation events
  Asymmetry | 465
  Biopsy | 17
  Breast - unacceptably high sensation | 2
  Breast pain not associated with other complication | 26
  Calcification | 1
  Capsular Contracture (Baker Grade II) | 238
  Capsular Contracture (Baker Grade III) | 423
  Capsular Contracture (Baker Grade IV) | 224
  Capsule / Pocket tear | 23
  Delayed wound healing | 37
  Extrusion | 90
  Granuloma | 2
  Hematoma | 128
  Hypertrophic scarring | 104
  Implant removal | 76
  Infection | 142
  Irritation / Inflammation | 12
  Lack of projection | 54
  Necrosis | 11
  New diagnosis of breast cancer | 17
  New diagnosis of rheumatic disease | 1
  Nipple - unacceptably low sensitivity | 2
  Nipple complications | 25
  Palpability - implant | 9
  Position change (dissatisfaction) | 313
  Ptosis | 128
  Rupture | 41
  Seroma | 33
  Size change - patient request | 624
  Size change - physician assessment only | 37
  Staged Reconstruction | 7
  Symmastia | 26
  Wrinkling | 76
  Unknown | 513
  Other | 139

ADVERSE EVENTS:
Description: In the Original study, follow-up data were to be collected by survey in years 1-10. Surgeons were also to see MemoryGel participants in years 1, 4-6, and 9-10. All local complications, reasons for reoperation, and reasons for removal reported by the participant or surgeon were to be recorded. In 2015 FDA approved a redesign of the study whereby data collection was limited to only reoperation data for MemoryGel participants and the reasons for reoperation. These are presented as Outcome Measures.
Groups:
- Overall Study: Subjects in either the MemoryGel group or the saline breast implant control group
Arm/Group | Overall Study
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The data presented may represent an under-estimation of reoperation and explantation rates due to the lack of mandatory safety reporting and ability for participants to be treated at non-study sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT00756652/Prot_SAP_000.pdf